CLINICAL TRIAL: NCT02149628
Title: The Effect of Propofol Based Total Intravenous Anesthesia on Oxidative Stress and Nitric Oxide in Patients Undergoing Laparoscopic Surgery
Brief Title: The Effect of Propofol Based Total Intravenous Anesthesia on Oxidative Stress and Nitric Oxide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2013-0098
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- desflurane (Active Comparator): use desflurane as a primary anesthetics during anesthesia guided by bispectral index (BIS)
  Interventions: Drug: Desflurane
- propofol (Experimental): propofol infusion with target-controlled infusion(TCI) device guided by BIS
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol
  Other Names: fresofol, 2%
  Arms: propofol
Drug: Desflurane
  Arms: desflurane

SUMMARY:
Robot assisted laparoscopic radical prostatectomy(Robot-LRP) requires pneumoperitoneum and trendelenburg position which result in oxidative stress and inflammatory response.

Propofol is well known to reduce those responses during anesthesia. Therefore, we try to figure out the efficacy of propofol to reduce oxidative stress, inflammatory response and increase the nitric oxide activity during robot-LRP compared to that of desflurane.

To investigate the oxidative stress, malondialdehyde will be measured. As inflammatory markers, interleukin-1β, interleukin-6, tumor necrosis factor-α will be measured. Nitric oxide will be measured as well.

Secondarily, kidney protection effect of propofol over desflurane will be compared.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing robot-assisted laparoscopic radical prostatectomy under general anesthesia

Exclusion Criteria:

* chronic renal failure ( estimated glomerular filtration rate <60 mL/min/1.73m2)
* allergy to propofol, nuts
* on diuretics, vitamin C or vitamin E within 5 days before surgery
* Body mass index > 30 kg/m2
* older than 70 years
* who cannot read the patient consent form

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
changes of serum malondialdehyde, Interleukin-1β, interleukin-6, tumor necrotic factor-α, nitric oxide during operation | 100 min after pneumoperitoneum, 10 min after decompression

SECONDARY OUTCOMES:
kidney function after anesthesia | 1 day after operation
  measure creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Goun Roh, MD, Principal Investigator — Yonsei University Gangnam Severance Hospital
Locations (1):
- Yonsei University, Gangnam Severance Hospital, Seoul, South Korea